CLINICAL TRIAL: NCT01362322
Title: Immunogenicity and Safety Study of GSK Biologicals' Boostrix™ Vaccine Using a New Syringe Presentation in Healthy Adolescents Aged 10-15 Years
Brief Title: Immunogenicity and Safety of BoostrixTM Using a New Syringe in 10 to 15-year Old Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 114778
Record Dates: First submitted 2011-05-19; First posted 2011-05-30 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-05

CONDITIONS: Diphtheria; Tetanus; Acellular Pertussis
Keywords: dTpa; Boostrix
MeSH Terms: conditions — Diphtheria; Tetanus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BOOSTRIX NEW GROUP (Experimental): Subjects, aged 10 to 15 years, received one dose of Boostrix™ vaccine administered using a new syringe presentation (prefilled syringes from a different manufacturer) in the deltoid of the non-dominant arm, at Day 0.
  Interventions: Biological: Boostrix TM (new syringe presentation)
- BOOSTRIX PREV GROUP (Active Comparator): Subjects, aged 10 to 15 years, received one dose of Boostrix™ vaccine administered using a previous syringe presentation (single dose vial or a prefilled disposable syringe without a needle) in the deltoid of the non-dominant arm, at Day 0.
  Interventions: Biological: Boostrix TM (previous syringe presentation)

INTERVENTIONS:
Biological: Boostrix TM (new syringe presentation) — Single dose, intramuscular administration in a new syringe presentation
  Arms: BOOSTRIX NEW GROUP
Biological: Boostrix TM (previous syringe presentation) — Single dose, intramuscular administration in previous syringe presentation
  Arms: BOOSTRIX PREV GROUP

SUMMARY:
The purpose of the study is to compare the immunogenicity and safety of a booster dose of BoostrixTM administered in a new syringe presentation to that of BoostrixTM administered in the previous syringe presentation in healthy adolescents aged 10-15 years.

DETAILED DESCRIPTION:
The protocol has been updated following Protocol amendment 1 date 03 August 2011 leading to the update of the exclusion criteria to allow subjects in Mexico to receive the flu vaccine in accordance with the local standard of care.

The protocol has been updated following Protocol amendment 2 dated 14 December 2011 due to the recruitment constraints as a result of the DT/dTpa vaccination campaign in the countries. The inclusion and exclusion criteria were amended to allow the participation of those who have already received the 6th dose of the diphtheria, tetanus and/or pertussis containing vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/Legally Acceptable Representative(s) and subjects who the investigator believes can and are willing to comply with the requirements of the protocol.
* A male or female between 10 and 15 years of age at the time of booster vaccination.
* Prior to protocol amendment 2, subjects who have previously received 5 doses of diphtheria-tetanus-pertussis vaccine (whole cell/acellular [w/a]) as part of primary and booster vaccination, in line with local recommendations.
* After protocol amendment 2, subjects who have previously received 6 doses of either DT(P) (w/a)/ dTpa vaccine as part of primary and booster vaccination, in line with local recommendations.
* Healthy subjects as determined by the investigator based on medical history and clinical examination before entering into the study.
* Written informed consent to be obtained before study entry from the parent(s)/ Legally Acceptable Representative(s) of the subject.
* Written informed assent to be obtained from the subject in addition to the informed consent signed by the parent(s)/ Legally Acceptable Representative(s), if required by local regulations.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has a negative pregnancy test on the day of vaccination,
  * if sexually active, has practiced adequate contraception for 30 days prior to vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after booster vaccination.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the booster dose of vaccine - with the exception of influenza vaccine which is allowed up to 7 days before the study vaccine dose, or planned in the period ≥ 7 days after the study vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* A history of previous or intercurrent diphtheria, tetanus or pertussis disease.
* A history of vaccination against these diseases since the 5th or the 6th dose of DT(P)/dT(pa). For subjects who have received the 6th dose of the diphtheria, tetanus and/or pertussis containing vaccine, the interval between the last DT(P)/dT(pa) vaccination and the administration of the study vaccine should be at least 18 months.
* Occurrence of any of the following adverse event after a previous administration of a Boostrix vaccine :

  * known hypersensitivity to any component of the vaccine, or have shown signs of hypersensitivity after previous administration of diphtheria, tetanus or pertussis vaccines,
  * encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine,
  * transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions, if applicable.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 671 (Actual)
Dates: Start 2011-07-01; Primary Completion 2012-09-03 (Actual); Study Completion 2012-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Santiago, Chile
- Mexico (2):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Estado de México

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pavia-Ruz N, Abarca K, Lepetic A, Cervantes-Apolinar MY, Hardt K, Jayadeva G, Kuriyakose S, Han HH, de la O M. Evaluation of a new syringe presentation of reduced-antigen content diphtheria, tetanus, and acellular pertussis vaccine in healthy adolescents--A single blind randomized trial. Hum Vaccin Immunother. 2015;11(7):1770-4. doi: 10.1080/21645515.2015.1041697. PMID 26075317
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Boostrix New Group | Boostrix Prev Group
Started | 335 | 336
Completed | 330 | 329
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix New Group | Boostrix Prev Group | Total
Number analyzed (Participants) | 335 | 336 | 671
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.9 (1.59) | 11.9 (1.61) | 11.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 178 | 357
  Male | 156 | 158 | 314

OUTCOME MEASURES:

1. Primary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: At Month 1
Population: The analysis was performed on the According To Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
IU/mL
  Anti-D | 6.784 [6.178 to 7.45] | 6.493 [5.915 to 7.128]
  Anti-T | 18.937 [17.313 to 20.713] | 18.515 [16.851 to 20.342]
Statistical Analysis 1: Comparison: Boostrix New Group vs Boostrix Prev Group; Analysis was performed to demonstrate that Boostrix administered using the new syringe presentation was non-inferior to Boostrix administered using the previous syringe presentation, in terms of immune response to diphteria vaccine antigens, one month after booster vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit (UL) of the 95% confidence interval (CI) on the geometric mean concentration (GMC) ratios [Boostrix-Prev Group over Boostrix-New Group] for anti-diphtheria (anti-D) antibodies was ≤ 1.5 (clinical limit for non-inferiority); ANCOVA; Adjusted radio = 0.96, 95% CI 2-sided [0.85 to 1.09]
Statistical Analysis 2: Comparison: Boostrix New Group vs Boostrix Prev Group; Analysis was performed to demonstrate that Boostrix administered using the new syringe presentation was non-inferior to Boostrix administered using the previous syringe presentation, in terms of immune response to tetanus vaccine antigens, one month after booster vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit (UL) of the 95% confidence interval (CI) on the geometric mean concentration (GMC) ratios [Boostrix-Prev Group over Boostrix-New Group] for anti-tetanus (anti-T) antibodies was ≤ 1.5 (clinical limit for non-inferiority); ANCOVA; Adjusted Ratio = 0.97, 95% CI 2-sided [0.86 to 1.1]

2. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter(EL.U/mL)
Time Frame: At Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
EL.U/mL
  Anti-PT: number analyzed (Participants) | 318 | 318
  Anti-PT | 140.2 [126 to 156.1] | 125.9 [112.7 to 140.7]
  Anti-FHA: number analyzed (Participants) | 319 | 319
  Anti-FHA | 1080.2 [995.2 to 1172.5] | 1013.7 [940 to 1093.2]
  Anti-PRN: number analyzed (Participants) | 321 | 318
  Anti-PRN | 652.4 [572.1 to 743.9] | 619.2 [546 to 702.2]
Statistical Analysis 1: Comparison: Boostrix New Group vs Boostrix Prev Group; Analysis was performed to demonstrate that Boostrix administered using the new syringe presentation was non-inferior to Boostrix administered using the previous syringe presentation, in terms of immune response to pertussis toxoid vaccine antigens, one month after booster vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit (UL) of the 95% confidence interval (CI) on the geometric mean concentration (GMC) ratios [Boostrix-Prev Group over Boostrix-New Group] for anti-pertussis toxoid (anti-PT) antibodies was ≤ 1.5 (clinical limit for non-inferiority); ANCOVA; Adjusted Ratio = 0.92, 95% CI 2-sided [0.82 to 1.04]
Statistical Analysis 2: Comparison: Boostrix New Group vs Boostrix Prev Group; Analysis was performed to demonstrate that Boostrix administered using the new syringe presentation was non-inferior to Boostrix administered using the previous syringe presentation, in terms of immune response to filamentous haemagglutinin vaccine antigens, one month after booster vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit (UL) of the 95% confidence interval (CI) on the geometric mean concentration (GMC) ratios [Boostrix-Prev Group over Boostrix-New Group] for anti-filamentous haemagglutinin (anti-FHA) antibodies was ≤ 1.5 (clinical limit for non-inferiority); Adjusted Ratio = 0.92, 95% CI 2-sided [0.83 to 1.03]
Statistical Analysis 3: Comparison: Boostrix New Group vs Boostrix Prev Group; Analysis was performed to demonstrate that Boostrix administered using the new syringe presentation was non-inferior to Boostrix administered using the previous syringe presentation, in terms of immune response to pertactin vaccine antigens, one month after booster vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit (UL) of the 95% confidence interval (CI) on the geometric mean concentration (GMC) ratios [Boostrix-Prev Group over Boostrix-New Group] for anti-pertactin (anti-PRN) antibodies was ≤ 1.5 (clinical limit for non-inferiority); Adjusted ratio = 0.98, 95% CI 2-sided [0.85 to 1.13]

3. Primary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: as for outcome 1
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
IU/mL
  Anti-D | 0.472 [0.403 to 0.553] | 0.456 [0.392 to 0.53]
  Anti-T | 0.956 [0.835 to 1.095] | 0.899 [0.789 to 1.026]

4. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
EL.U/mL
  Anti-PT PRE: number analyzed (Participants) | 320 | 319
  Anti-PT PRE | 7.5 [6.6 to 8.7] | 7.2 [6.3 to 8.2]
  Anti-FHA PRE: number analyzed (Participants) | 316 | 315
  Anti-FHA PRE | 48.9 [43.3 to 55.2] | 49.4 [43.6 to 56]
  Anti-PRN PRE | 14 [12.3 to 15.9] | 13.4 [11.9 to 15]

5. Secondary Outcome: Number of Seropositive Subjects Against Diphtheria (D) and Tetanus (T) Antigens
Description: A seroprotected subject was defined as a subject whose antibody concentration was greater than or equal to (≥) 0.1. international units per milliliter (IU/mL), as assessed by the Enzyme Linked Immunosorbent Assay (ELISA).
Time Frame: At Day 0 (PRE) and at Month 1 (POST)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
Participants
  Anti-D PRE | 284 | 286
  Anti-D POST | 320 | 319
  Anti-T PRE | 311 | 314
  Anti-T POST | 321 | 319

6. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Antigens
Description: A seroprotected subject is defined as a vaccinated subject with anti-D and anti-T antibody concentration greater than or equal to ( ≥) 1 international units per milliliter (IU/mL).
Time Frame: At Day 0 (PRE) vaccine and at Month 1 (POST)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
Participants
  Anti-D PRE | 83 | 89
  Anti-D POST | 315 | 310
  Anti-T PRE | 151 | 143
  Anti-T POST | 321 | 319

7. Secondary Outcome: Number of Seropositive Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations)
Description: A seroprotected subject was defined as a subject whose antibody concentration was greater than or equal to (≥) 5 Enzyme Linked Immunosorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Day 0 (PRE) vaccine and at Month 1 (POST)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
Participants
  Anti-PT PRE: number analyzed (Participants) | 320 | 319
  Anti-PT PRE | 175 | 175
  Anti-PT POST: number analyzed (Participants) | 318 | 318
  Anti-PT POST | 316 | 315
  Anti-FHA PRE: number analyzed (Participants) | 316 | 315
  Anti-FHA PRE | 310 | 310
  Anti-FHA POST: number analyzed (Participants) | 319 | 319
  Anti-FHA POST | 319 | 319
  Anti-PRN PRE | 269 | 272
  Anti-PRN POST: number analyzed (Participants) | 321 | 318
  Anti-PRN POST | 321 | 318

8. Secondary Outcome: Number of Subjects With Booster Response to Diphtheria (D) and Tetanus (T) Antibodies
Description: Booster response to the diphtheria and tetanus antigens, was defined as: for initially seronegative subjects (pre-vaccination concentration <0.1 IU/mL): antibody concentrations at least 4 times the cut-off (post-vaccination concentration ≥ 0.4 IU/mL); for initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least 4 times the pre-vaccination concentration.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 319
Participants
  Anti-D | 257 | 252
  Anti-T | 266 | 270

9. Secondary Outcome: Number of Subjects With a Booster Response to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA), Pertactin (PRN) Antigens.
Description: Booster response to the PT, FHA and PRN antigens, was defined as: for initially seronegative subjects: antibody concentrations at least 4 times the cut-off (post-vaccination concentration ≥ 20 EL.U/mL); for initially seropositive subjects with pre-vaccination concentration ≥ 5 EL.U/mL and < 20 EL.U/mL: an increase in antibody concentrations of at least 4 times the pre-vaccination concentration; and for initially seropositive subjects with pre-vaccination concentration ≥ 20 EL.U/mL: an increase in antibody concentrations of at least 2 times the pre-vaccination concentration.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 321 | 318
Participants
  Anti-PT: number analyzed (Participants) | 317 | 318
  Anti-PT | 298 | 295
  Anti-FHA: number analyzed (Participants) | 314 | 315
  Anti-FHA | 305 | 304
  Anti-PRN | 315 | 317

10. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 4 days (Days 0-3) post vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with documented administration of the study vaccine and with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 330 | 329
Participants
  Any Pain | 237 | 248
  Any Redness | 113 | 94
  Any Swelling | 98 | 90

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Days 0-30) post
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with documented administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 335 | 336
Participants | 44 | 45

12. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache and gastrointestinal symptoms. Gastrointestinal symptoms included Nausea, Vomiting, Diarrhea and or Abdominal pain. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 4 days (Days 0-3) post vaccination period
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 330 | 329
Participants
  Any Fatigue | 83 | 86
  Any Gastrointestinal symptoms | 32 | 42
  Any Headache | 88 | 108
  Any Temperature | 9 | 6

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0 - Month 1)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix New Group | Boostrix Prev Group
Number analyzed (Participants) | 335 | 336
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms during the 4-day post-vaccination period (Day 0 - Day 3), Unsolicited AEs during the 31-day post-vaccination period (Day 0 - Day 30), SAEs during the entire period (Day 0 - Month 1).
Arm/Group | Boostrix New Group | Boostrix Prev Group
Serious Adverse Events (participants affected / at risk) | 1/335 | 0/336
Other Adverse Events (participants affected / at risk) | 263/335 | 279/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix New Group (N=335) | Boostrix Prev Group (N=336)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix New Group (N=335) | Boostrix Prev Group (N=336)
Erythema (Skin and subcutaneous tissue disorders) | 113 (113) | 94 (94)
Fatigue (General disorders) | 83 (83) | 86 (86)
Gastrointestinal disorder (Gastrointestinal disorders) | 32 (32) | 42 (42)
Headache (Nervous system disorders) | 89 (90) | 109 (110)
Pain (General disorders) | 237 (237) | 248 (248)
Swelling (General disorders) | 98 (98) | 90 (90)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.